CLINICAL TRIAL: NCT02347514
Title: Implementing Diabetes Group Visits in Community Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB14-0973
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes Group Visit (Experimental): Subjects in this arm will be asked to attend one group visit at their health center each month for six months. The group visits will involve various staff and providers at the health center who will teach them how to take care of their diabetes. Subjects will be scheduled to attend the same group visit appointments as the other subjects, and health center staff will encourage the group to share their own experiences about living with diabetes with the rest of the group.
  If subjects at the health center additionally implementing the text-messaging intervention consent to enroll in the study, their phone number will also be entered into a secure system that will allow the group visit healthcare team to send them text messages during the course of the six months they are in the program. These text messages are intended to offer the subjects additional support in taking care of their diabetes.
  Interventions: Behavioral: Diabetes group visit
- Usual care (No Intervention): Patients in the control arm will be selected after the follow-up period is over for the intervention arm. They will receive the care they normally receive at their health center.

INTERVENTIONS:
Behavioral: Diabetes group visit
  Arms: Diabetes Group Visit

SUMMARY:
Community health centers across the US are seeking to address the growing prevalence of diabetes in adults. The University of Chicago has partnered with the MidWest Clinicians' Network (MWCN) to conduct a research study to train community health center staff and providers to implement and sustain diabetes group visits, also referred to as shared medical appointments, at their health center. The study's aims are to: 1) Develop, conduct, and evaluate a training program for health center staff to implement a diabetes group visit intervention in their health center; 2) Assess the implementation of diabetes group visits in the community health center setting and determine the cost of implementation; 3) Assess the feasibility and cost of implementing a text-messaging intervention in addition to the implementation of diabetes group visits in the CHC setting at one health center and 4) Assess the impact of the diabetes group visits alone and diabetes group visits plus text-messaging on diabetes process measures, patient outcomes, and patient satisfaction compared to control patients from the same health center with six months of follow-up once the six-month group visit program ends.

DETAILED DESCRIPTION:
Community health centers across the US are seeking to address the growing prevalence of diabetes in adults. The University of Chicago has partnered with the MidWest Clinicians' Network (MWCN) to conduct a research study to train community health center staff and providers to implement and sustain diabetes group visits, also referred to as shared medical appointments, at their health center. The study's aims are to: 1) Develop, conduct, and evaluate a training program for health center staff to implement a diabetes group visit intervention in their health center; 2) Assess the implementation of diabetes group visits in the community health center setting and determine the cost of implementation; 3) Assess the feasibility and cost of implementing a text-messaging intervention in addition to the implementation of diabetes group visits in the CHC setting at one health center and 4) Assess the impact of the diabetes group visits alone and diabetes group visits plus text-messaging on diabetes process measures, patient outcomes, and patient satisfaction compared to control patients from the same health center with six months of follow-up once the six-month group visit program ends.

The MWCN Research Committee is looking for six community health center (CHC) teams comprised of three to four members to participate in the study. The study will last 18 months and will require study participants to complete the following activities as part of the study:

* Attend two mandatory learning sessions in Chicago in the spring and fall of 2015 that will each last two days (Friday and Saturday all day, 9am-5pm)
* Participate in a mandatory third learning session conducted through a series of 4 or 5 weekly webinars in the spring of 2016
* Participate in monthly conference calls and/or webinars intended for tracking progress, trouble-shooting obstacles encountered, and further training in the months between each learning session
* Complete a training in the protection of human subjects in research
* Implement a monthly diabetes group visit intervention for at least six months at their health center
* Recruit 15 health center patients with diabetes who might benefit from participating in diabetes group visits to enroll in the program
* Complete four surveys (20-60 minutes each), one brief evaluation (10-15 minutes), monthly time and expense logs, and one telephone interview (25-40 minutes) between February 2015 and May 2016
* Collect patient data through survey administration at two time-points for patients who attend at least one group visit session and through telephone interviews for 1) patients who said they would enroll in the group visit program but who did not attend at least one session and 2) patients who attended less than four group visit sessions
* Collect patient data through EMR / chart abstraction for up to 15 patients who enroll in the group visit program at three study time points over the course of a year from mid-2015 to mid-2016 and for up to 30 patients who do not participate in the group visit program and who will serve as control patients for the study.at one point in mid-2016.

The learning sessions will include various module topics that have been developed based on a review of the current literature of diabetes group visit interventions, preliminary research done through site visits to CHCs with diabetes group visit experience, and input from the MWCN Research Committee. The learning sessions will also provide the opportunity for each health center to share their own unique experiences and to learn from other health centers' experiences.

The first learning session will provide an overview of the benefits of group visits, "best practices" for implementing a diabetes group visit program in a health center, the barriers and challenges that may arise in implementing diabetes group visits, strategies to overcome these barriers, and factors that facilitate the implementation of group visits and affect their sustainability. During the first learning session, participating health centers will also have some time to develop a detailed plan for the implementation of a group visit program at their center. In addition, they will learn how to evaluate the implementation of their program and the impact of their program on patient outcomes. Each team will also be given a patient curriculum guide which they can tailor to the needs of their patient population and use to implement the diabetes group visit program in their health center. The health center selected to implement the text-messaging intervention in addition to the group visit intervention will be asked to attend additional training modules relating to the implementation of the text-messaging intervention.

During the six months following the first learning session, each health center will implement their individualized program implementation plan, using rapid "Plan-Do-Study-Act" quality improvement strategies to design, implement and evaluate their program. Ongoing conference call meetings, webinars and listserv communications will provide additional opportunities for sharing, problem solving, and peer support. The second learning session will occur after approximately six months, and is designed to allow CHC group visit teams to present de-identified and aggregated baseline group visit patient data and discuss any obstacles or challenges that they have encountered thus far. The third learning session will be held a year after the first session, during which time CHC group visit teams will present their six-month de-identified and aggregated group visit patient data, describe how they have overcame challenges that arose throughout implementation, and discuss concerns regarding sustainability. These team presentations will take place online via hour-long webinars that will take place each week for approximately one month.

This collaborative effort will employ a standard method of data collection across participating health centers to assess CHC provider/staff training participant satisfaction with the training, their perceived utility and acceptability of the training, as well as their confidence in being able to implement and sustain a group visit program in their health center. Process outcomes will include the number of group visit sessions held; attendance rates; program costs; and challenges, barriers, facilitators and benefits identified during the process of implementing the group visits. Patient level data (A1c, blood pressure, BMI, self-care behaviors, satisfaction) will also be collected and analyzed to explore possible effects of the group visit intervention on patient outcomes.

Expected products from this project include an evaluation of the training and the group visit intervention implemented in six Midwestern community health centers, the dissemination of best practices for implementing diabetes group visits in the community health center setting, and the subsequent development of this pilot program into a full scale randomized controlled trial across multiple community health centers. This pilot study will also help participating health centers problem-solve in order to overcome challenges in implementing and sustaining programs at their health center and understand how to provide better care to their patients in the areas of behavior modification and diabetes management. Finally the pilot conducted at the center selected to implement the text-messaging intervention in addition to the group visit intervention will provide information of the feasibility of additionally implementing a text-messaging intervention and explore whether such a combined intervention could have the potential to improve attendance at group visit appointments, change health behavior, and improve patient outcomes to a greater extent than group visits alone.

Application Requirements:

Health centers interested in applying to participate in this research study will be expected to:

* Contact the study coordinator to be screened for eligibility before completing the application.
* Complete the attached application and submit it by the specified deadline along with letters of support from both the Executive Director / CEO and the Medical Director of the health center stating their endorsement and support for the participation of their center's staff in this QI training and program implementation initiative.
* Designate a minimum of three to four staff/providers at their center who will fully participate in the study's activities as described on the first page of this request for applications.
* Agree to collect and report the de-identified group visit patient baseline, 6-month and 12-month data and the post-follow-up period control patient data listed in the application through EMR / chart abstraction, as well as, collect and report additional de-identified patient data through survey administration and select telephone interviews.

The MWCN Research Committee will review all applications and select the six health centers that represent different regions of the Midwest, offer a diverse set of patient populations, and demonstrate the greatest interest in and ability to attend the learning sessions, implement the diabetes group visit program at their center, and collaborate in the evaluation of the training and group visit intervention. If selected to participate in the study, the health center's executive director / CEO and medical director will be asked to sign an enrollment contract acknowledging the requirements of the study and stating they will support the group visit team of three to four staff and providers in completing the study requirements.

Health center recruitment for this study has closed. Recruitment of patients within selected health centers will start in May 2015.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Patients must have been a patient at the health center since the beginning of 2013
* Patients must have attended at least two appointments at the health center within the past year
* Patients must have a diagnosis of type 2 diabetes
* (For group visit patients only) Patients' last documented A1c result must have been greater than or equal to 8.0% and the test must have been done during the last 18 months at the time of the selection
* (For group visit plus text-messaging patients only) Patients must own a cellular phone with text-messaging capabilities
* (For control patients only) Patients must have attended at least three individual appointments at the health center between February 2015 and July 2016.
* (For control patients only) Patients' last documented A1c result prior to the start of the group visit program must have been greater than or equal to 8.0% and the test must have been done during the 18 months prior to the start of the group visit program

Exclusion Criteria:

Patients who are under 18 years old, have not been a patient at the health center since the beginning of 2013, have not attended at least two appointments at the health center within the past year, do not have a diagnosis of type 2 diabetes, have not had an A1c test done during the 18 months prior to the start of the group visit program, or whose last documented A1c result before the start of the group visit program was less than 8.0%, will be excluded from the study.

Pregnant women; patients with an uncontrolled psychiatric problem, such as schizophrenia, psychosis, dementia, or another cognitive impairment; and patients with hearing difficulties or a severe physical disability will also be excluded from the study.

Additionally, patients who do not own a cellular phone with texting capabilities will not be eligible for inclusion as an intervention patient subject at the group visit plus text-messaging health center site.

Patients who have not attended at least three individual appointments at the health center between February 2015 and July 2016 will not be eligible for inclusion as a control patient subject in the study.

Patients will also be excluded from participation in the study if their primary care provider deems they would not benefit from participation in a diabetes group visit program and/or does not provide approval for them to be in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-11; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
glycosylated hemoglobin | change from baseline to 6 months and 12 months.

SECONDARY OUTCOMES:
Summary of Diabetes Self-Care Activities (SDSCA) | change from baseline to 6 months and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States